CLINICAL TRIAL: NCT04324437
Title: eRAPID: Electronic Monitoring of Patient-reported Symptoms in Patients With a Diagnosis of Thoracic Cancer Managed at Leeds Cancer Centre
Brief Title: eRAPID: Online Symptom Reporting in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); Iqvia Pty Ltd (Industry)
Responsible Party: Principal Investigator, Galina Velikova, Professor, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 270042
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Thoracic Cancer; Non-small Cell Lung Cancer; Small-cell Lung Cancer; Pleural Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Mesothelioma, Malignant

STUDY DESIGN:
Intervention Model Description: Consecutive recruitment based on patient choice into two cohorts: access to internet at home or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eRAPID online symptom monitoring in lung cancer (Other): Two groups of patients with differing internet access: access from home or access in clinic only
  Interventions: Other: eRAPID online symptom monitoring in lung cancer

INTERVENTIONS:
Other: eRAPID online symptom monitoring in lung cancer — The eRAPID in lung cancer intervention is an online symptom monitoring system which provides tailored advice depending on the severity of symptoms reported. The system is integrated into the electronic medical record and results can be viewed by the medical team.

SUMMARY:
Lung cancer is a leading cause of cancer-related ill-health and death in the United Kingdom (UK), but with advances in systemic anti-cancer therapies the prognosis for people in later stages is improving. There is growing evidence that electronic systems which enable patients to monitor and report symptoms can help improve symptom control and patient care. This study aims to investigate optimal ways of introducing an electronic symptom reporting system (eRAPID) in lung cancer care at Leeds Cancer Centre. eRAPID was developed by the University of Leeds and its integration with the electronic health records at Leeds Cancer Centre enables staff to view patient symptom reports directly. eRAPID provides advice to patients about self-management of milder symptoms, for serious symptoms patients are encouraged to contact the hospital and an alert is sent to the nurse or doctor by email.

The aim of the study is to assess the feasibility and usefulness of an electronic symptom reporting system (eRAPID) for lung cancer patients and healthcare professionals during the treatment of lung cancer and during one year follow up.

Two groups of patients will be recruited on the basis of their access to the internet at home (rather than randomisation). It is anticipated that approximately 100 patients will enrol into one of two groups:

* Group 1: Patients with online access at home will be asked to report weekly using their own devices.
* Group 2: Patients without online access will be asked to report on a tablet computer before their planned clinic appointments.

The eRAPID questionnaire is based on existing eRAPID items with the addition of new items specific to lung cancer. These have been developed by the clinical team and patient groups have been consulted over the suitability of the wording used.

Analysis of patient reported symptoms, quality of life and clinical information will be descriptive. Disease-related symptoms and health-related quality of life will be compared across groups of patients with a diagnosis of lung cancer. Treatment-related side effects of patients will be compared across the different types of treatment received. To determine the best means of engaging patients in systematic electronic reporting, the recruitment and compliance rate will be compared between the two patient groups. The utility of patient reported information to healthcare staff will be assessed through staff interviews.

DETAILED DESCRIPTION:
Background: Lung cancer is a leading cause of cancer-related morbidity and mortality. There are 2 main categories of lung cancer: non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC). NSCLC accounts for approximately 85% of lung cancer diagnoses, almost 70% of NSCLC cases are diagnosed in the advanced/metastatic stages (IIIB-IV) of the disease. Pleural mesothelioma is another rare form of lung cancer, the average incidence across European countries is 20 cases per million people. Historically, patients with NSCLC were treated with the same algorithm, without consideration of their histological sub-type or their molecular profile. More recently, personalised therapies based on histology and/or molecular pathology have become the standard of care. The stage of NSCLC determines treatment options, with surgery being the mainstay of treatment for patients in early stages of the disease (stages I-IIIA). Additionally, those with localised disease spread (stages II and IIIA) may receive adjuvant therapy [11]. In patients with advanced/metastatic disease (stages IIIB-IV) and a performance status (PS) score of 0-2, the first line treatment options include chemotherapy regimens with or without immunotherapy or targeted biological therapy.

Patient reported outcome measures (PROMs) encompass data self-reported by patients about how they feel and function and include symptoms, physical function, emotional distress and health-related quality of life (HRQoL). PROMs are becoming important for patient care, as they provide the means of recording the experience of the patient in a structured format readily available to relevant clinical staff. Recently a randomised control trial (RCT) in advanced lung cancer using web-mediated follow-up showed overall survival benefit of 7-9 months compared to usual care, whilst maintaining cost-effectiveness. The relapses were detected earlier in patients in the intervention arm facilitating earlier and appropriate treatment initiation compared to patients in the control arm.

Study aims: This study will systematically capture patient reported disease-related symptoms, treatment-related side effects and HRQoL in a cohort of patients treated with systemic anti-cancer therapy (SACT) for thoracic cancer. The objectives are:

1. To compare disease-related symptoms and HRQoL across groups of patients stratified by patient and clinical characteristics.
2. To compare treatment-related side effects of patients prescribed chemotherapy, tyrosine kinase inhibitors (TKIs) or checkpoint inhibitors.
3. To compare outcomes, such as healthcare resource utilisation (HCRU), in patients systematically self-reporting symptoms
4. To examine patient acceptance, feasibility of this approach and optimal means of engaging with patients in the systematic PROMs reporting in a real world setting.
5. To assess the utility of PROMs reported by patients to their healthcare professionals.

Study design: This is an interventional, prospective study conducted at a single cancer centre. Patients with a diagnosis of thoracic cancer prescribed SACT will be enrolled in the study at oncology clinic visits. The intervention is an electronic patient self-report of disease-related symptoms, treatment-related side effects and HRQoL. This design allows the assessment of the utility to clinicians of PROMs reporting in the real world setting and provides an opportunity to study customised patient interventions based on PROMs reporting.

There will be two cohorts of patients. Cohort 1: Patients with online access at home, able to report PROMs from a location of their choice, using their own devices (laptop, tablet, smart phone). They will be requested to report weekly.

1. Cohort 2: Patients without online access who will complete PROMs on a tablet before their scheduled clinic appointment in a private space at Leeds Cancer Centre (LCC). Reporting frequency will be governed by frequency of routine clinical visits.

Table 1: SACT prescribed for enrollment in the study Diagnosis Treatment description

NSCLC Platinum-based chemotherapy:

* Carboplatin-based
* Cisplatin-based Non-platinum-based chemotherapy
* Pemetrexed TKIs Immune-checkpoint inhibitors (inc. anti-PDL1)

SCLC Platinum-based chemotherapy:

* Carboplatin-based
* Cisplatin-based Non-platinum-based chemotherapy

Pleural mesothelioma Platinum-based chemotherapy:

* Carboplatin-based
* Cisplatin-based Non-platinum-based chemotherapy
* Pemetrexed

Number of patients: All patients meeting patient selection criteria during the recruitment period will be invited to participate. Approximately 100 patients are expected to be enrolled (70 patients with a diagnosis of NSCLC, 20 patients with a diagnosis of SCLC, and 10 patients with a diagnosis of pleural mesothelioma). This estimation is based on the number of thoracic cancer patients receiving SACT at LCC, the proportion who relapse, and 75% of eligible patients enrolling.

Recruitment and study duration: Index date is defined in both cohorts as the initiation of a line of SACT within the study period. For patients newly diagnosed within the study period, this will be the initiation of their 1st line of therapy (LoT). For patients diagnosed prior to the study period, the index date will be initiation of 1st or subsequent LoT. Collecting baseline PROMs at the start of a LoT allows the analysis of change from baseline in disease- and treatment-related side effects with each new LoT. If the patient wishes to be enrolled, they will be trained how to use the system. The formal consent will be completed electronically and then participant complete baseline questionnaires on the electronic platform. Recruitment will occur over 12-months with 12-month follow-up. There will be an interim study review to assess the number of patients enrolled, description of patients enrolled, systematic PROMs reporting compliance, and interim participant feedback.

Instruments' reporting frequency: Three instruments will be used:

1. eRAPID Patient reported adverse events (PRAE) CTCAE adapted symptom questionnaire for lung cancer, including disease-related symptoms and treatment-related side effects
2. EORTC Quality of Life Questionnaire (QLQ-C30)
3. EuroQol General Quality of Life questionnaire Cohort 1 Patients (Online access) symptom questionnaire is to be completed weekly, and the quality of life questionnaires at baseline and then every 12 weeks over the year.

Cohort 2 Patients' (In clinic access) symptom questionnaire to be completed online before routine clinic appointment. Type of treatment and frequency of clinics will determine the frequency of questionnaire completion.

Software: eRAPID uses a web-based questionnaire builder system (QTool) to support the collection and clinical integration of patients' reports. Algorithmic questionnaire scoring generates severity-dependent management advice to patients and staff when patients self-reports using the PRAE CTCAE:

* Patients login to QTool using a unique user name and password, complete the questionnaires remotely on computers/mobile phones/tablets or on a tablet provided in clinic at LCC.
* Immediate, tailored advice derived from a series of algorithms is generated in response to reported symptoms and toxicities.
* If severe symptoms are reported, patients are advised to contact the hospital immediately and an alert is sent to a member of the clinical team.
* For mild/moderate complications, information about self-managing these issues are provided in QTool and hyperlinks to more detailed advice on the eRAPID patient websites.
* PROMs are available for patients to view in their QTool login and for clinicians to review in the individuals' electronic medical record.

Healthcare professionals' and patient feedback: Interviews will be conducted with healthcare professionals and patients about their views of using the eRAPID system. Five members of staff will be interviewed (n=3 oncologists, n=2 nurses) twice during the study period to gain feedback on the usefulness of the eRAPID system in lung cancer care. Approximately 12 patients will be interviewed at different stages of using the system from home or from clinic.

Clinical variables: Patient characteristics, clinical characteristics, treatment variables will be captured either prospectively in a study case report form (CRF) or retrospectively by extracting the data from hospital electronic systems.

Data analysis Baseline demographic and clinical data will be tabulated using frequencies and summary by age, gender, cancer pathology type, stage and treatments.

Recruitment strategy feasibility will be evaluated by summarising the eligibility and consent processes. The proportion of patients who meet the eligibility criteria in terms of cancer site, treatment type and timescale will be reported using information from the electronic health record. The number of patients completing the adverse events (AE) online vs those in clinic will be summarised. Where available, reasons for ineligibility and non-participation in the study will be summarised. Retention during the study, including the number of participants withdrawing from the study and the timing of and reasons for withdrawal will also be presented. The number of participants involved at each stage will be summarised (patients identified, approached, consented, completed symptoms and side effects).

The integrity of systems will be assessed by exploring any technical issues encountered during the study, summarising the rates of questionnaires not being fully completed (assessed by incomplete calls or time-outs depending on the system used). Reasons for patients completing symptoms and side effects in clinic rather than from home will be presented. Time taken to complete the questionnaires will be summarised using time stamps of start and end of calls/online sessions.

The numbers of expected and additional AE reports and severe AE alerts generated will be summarised overall, by cancer type, treatment and completion modality (online vs clinic). The number of telephone calls to hospital staff, acute admissions, ward stays, contacts with general practitioner and/or community services (where available) and number of deaths will be summarised overall and by treatment modality. Changes to supportive medication, treatment (chemotherapy, immunotherapy, targeted therapies) doses and treatment plans and the percentage of planned therapy received will be summarised overall and by treatment modalities. Differences between treatments may be explored using logistic or linear regression (as appropriate) adjusted for stratification factors. Clinician/staff acceptability will be explored by content analysis of the interviews and field notes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thoracic cancer: Non-small cell lung cancer (NSCLC), or Small cell lung cancer (SCLC), or Pleural mesothelioma
* Start of a systemic anti-cancer therapy with prescribed chemotherapy, tyrosine kinase inhibitors (TKIs) or checkpoint inhibitors within the recruitment period
* Willing and able to provide written informed consent
* Fluency in English

Exclusion Criteria:

* Cognitive impairment
* Receiving best-supportive care only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited/number of patients approached (consent rate) | Baseline
  Number of patients approached and recruited will be logged during recruitment
Number of participant withdrawals | 12 months
  Number of participant withdrawals will be logged at the time of withdrawal
Reason for participant withdrawal | 12 months
  Reasons for withdrawal will be captured in CRF at time of withdrawal
Use of the intervention | 6 month and 12 months
  Number of self-reported symptom monitoring reports and quality of life questionnaires completed
Acceptability of intervention to patients | 6 months and 12 months
  Interim and end of study interviews with patients
Acceptability of intervention to clinicians | 6 months and 12 months
  Interim and end of study interviews with clinicians
Integrity of the system | 6 months and 12 months
  Technical issues logged during the study
Proportion of missing data in symptom reports and quality of life questionnaires | 12 months
  Regular completions of symptom reports (either weekly or per scheduled clinical and quality of life questionnaires completed 12 weekly by participants
Number of adverse event reports, severe adverse event alerts and patient deaths | 12 months
  Descriptive statistics by cancer type, treatment and completion modality
Use of hospital services (triage calls, acute admissions, ward stays) | 12 months
  Descriptive statistics overall and completion modality
Changes to supportive medication, treatment doses and planned therapy | 12 months
  Descriptive statistics overall and completion modality

CONTACTS AND LOCATIONS:
Overall Officials: Galina Velikova, Principal Investigator — University of Leeds
Locations (1):
- St James's University Hospital, Leeds Teaching Hospital Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research group website and webpage relating to the study — https://pcor.org.uk/erapid-electronic-monitoring-of-patient-reported-symptoms-in-patients-with-a-diagnosis-of-thoracic-cancer-managed-at-leeds-cancer-centre/